CLINICAL TRIAL: NCT05458206
Title: Effect of Mulligan Snag and Diaphragmatic Release on Thoracic Kyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam omran Grase, lecturer at basic science department, faculty of physical therapy cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003548
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2022-11

CONDITIONS: Postural Kyphosis, Cervicothoracic Region

STUDY DESIGN:
Intervention Model Description: EFFECT OF MULLIGAN SNAG MOBILISATION AND DIAPHRAGMATIC RELEASE
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- diaphragmatic release, and conventional (Experimental): Diaphragmatic release:
  The patients will be positioned in the supine position. The therapist stood at the head of the patient. The therapist makes manual contact bilaterally under the costal cartilages of the lower ribs (7th to 10th ) with hypothenar regions of the hands and the last three fingers. During the patient's inspiration, the therapist will gently pull the points of hand contacts toward the head and slightly laterally, while elevating the ribs simultaneously. During exhalation, the therapist will deepen hand contact toward the inner coastal margins for 5 to 7 minute conventional therapy: the patient will receive chin-in, interscapular exercises, and pectoralis stretch
  Interventions: Other: mulligan snag mobilization and diaphragmatic release
- mulligan SNAG mobilization, and conventional (Experimental): mulligan snag: Apply a passive intervertebral movement in a superior anterior direction along the facet plane. While maintaining this "glide" as the patient actively moves in any range of physiological movement and then sustains it at the end range position for a few seconds. (3 sets,10 repetitions) conventional therapy: the patient will receive chin-in, interscapular exercises, and pectoralis stretch
  Interventions: Other: mulligan snag mobilization and diaphragmatic release
- mulligan SNAG mobilization, diaphragmatic release, and conventional (Experimental): Diaphragmatic release:
  The patients will be positioned in the supine position. The therapist stood at the head of the patient. The therapist makes manual contact bilaterally under the costal cartilages of the lower ribs (7th to 10th ) with hypothenar regions of the hands and the last three fingers. During the patient's inspiration, the therapist will gently pull the points of hand contacts toward the head and slightly laterally, while elevating the ribs simultaneously. During exhalation, the therapist will deepen hand contact toward the inner coastal margins. (5 to 7 minutes) mulligan snag: Apply a passive intervertebral movement in a superior anterior direction along the facet plane. While maintaining this "glide" as the patient actively moves in any range of physiological movement and then sustains it at the end range position for a few seconds(3 sets,10 repetitions) conventional therapy: the patient will receive chin-in, interscapular exercises, and pectoralis stretch
  Interventions: Other: mulligan snag mobilization and diaphragmatic release
- the conventional therapy (Active Comparator): the patient will receive chin-in, inter-scapular exercises, and pectoralis stretch (3 sets,10 repetitions)
  Interventions: Other: mulligan snag mobilization and diaphragmatic release

INTERVENTIONS:
Other: mulligan snag mobilization and diaphragmatic release — The patients will be in the supine position. The therapist makes manual contact bilaterally under the costal cartilages of the lower ribs (7th to 10th ). During the patient's inspiration, the therapist will gently pull the points of hand contacts toward the head and slightly laterally. During exhalation, the therapist will deepen hand contact toward the inner coastal margins.
  mulligan snag, Apply a passive intervertebral movement in a superior anterior direction along the facet plane. While maintaining this "glide" as the patient actively moves in any range of physiological movement

SUMMARY:
the aim of this study is to investigate the efficacy of mulligan snag mobilisation and diaphragmatic release on upper crossed syndrome

DETAILED DESCRIPTION:
Acquired postural disorders can be a consequence, to a large extent, of contemporary living and working conditions. Some of the most typical factors include continuous use of mobile phones and computers, working in sedentary jobs. Prolonged incorrect posture and reduced physical activity present a dis-balance in the musculature . It can also lead to vision issues, as well as headaches, musculoskeletal issues, and pain, as well as a multitude of other symptoms.

Upon the available research studies, there is not study conducted to investigate the effect of mulligan SNAG mobilization and diaphragmatic release in upper crossed syndrome patients this trial has four groups; one will receive diaphragmatic release + conventional, the second will receive mulligan SNAG mobilization, and conventional, the third will receive mulligan SNAG mobilization+diaphragmatic release+conventional, the fourth subjects will receive conventional

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 17 to 22 years .
* Body Mass Index from 20 to 25 kg/m² .
* All participants have an intensity of neck pain on VAS (4-8) (moderate cases) .
* The subjects were chosen from both sexes.
* All participants have kyphosis angle ≥42°
* All participants have mechanical neck pain and FHP (craniovertebral angle CVA < 49) CVA of < 49) .

Exclusion Criteria:

* Malignancy
* Fractures of the cervical spine
* Cervical radiculopathy or myelopathy
* Vascular syndromes such as vertebrobasilar insufficiency
* Rheumatoid arthritis
* Neck or upper back surgery
* Taking anticoagulants
* Local infection
* Whiplash injury

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  The scale that will be used is the Visual analogue scale;each subject will be instructed to put point on a line from no pain to tolerable pain

SECONDARY OUTCOMES:
cervical range of motion | up to four weeks
  theCROM device will placed on patient's head while he/she seated and looking forward the difference between the ponter value and the value after movement will be recorded as the motion angle of the cervical vertebrae

OTHER OUTCOMES:
forward head | up to four weeks
  the craniovertebral angle (CVA) (the angle between the horizontal lines passing through and a line extending from the tragus of the ear to C7 notably). Lesser CVA indicates greater FHP
kyphotic angle | up to four weeks
  the bubble inclinometer is gravity-dependent, it is first zeroed on a vertical wall prior to measurement. Using a standard clinical procedure. the cephalic foot of the inclinometer will be placed on the pencil mark already on the C7 spinous process. This procedure will be repeated for the lower thoracic spine, with the caudal foot of the inclinometer placed on the pencil mark for T12. Both inclinometer angles will be recorded, taking care to minimize parallax error with each measurement by ensuring the recorder's eyes are on the same horizontal plane as the inclinometer. The thoracic kyphosis measure from the inclinometer readings will be obtained by taking the difference between the two measurements.
chest expansion | up to four weeks
  Measurements will be taken with the participants in a standing position with their arms along the body. The physiotherapist placed the "0" of the cloth tape measure on the appropriate vertebrae. The cloth tape will be held with an index finger between the participant's body and the cloth tape, without generating any deformation or cutaneous folds. The inspiratory diameter will be subtracted from the expiratory diameter to calculate the CE value.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of physical therapy Cairo university, Cairo, Giza Governorate
  - Faculty of physical therapy, Cairo, Giza Governorate